CLINICAL TRIAL: NCT03925207
Title: Retrobulbar Block and/or General Anesthesia for Orbital Ball Implants After Enucleation Surgery.: a Retrospective Observational Study
Brief Title: Retrobulbar Block and/or General Anesthesia for Orbital Ball Implants After Enucleation Surgery.
Acronym: pprb
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-2-18
Record Dates: First submitted 2019-02-26; First posted 2019-04-24 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Enucleated; Eye
Keywords: retrobulbar block; general anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrobulbar block is used to provide perioperative analgesia and anesthesia for orbital ball implants after enucleation surgery in the investigator's hospital. Retrobulbar block alone can provide quicker recovery, decreased time to discharge, opioid sparing, reduced costs. However, patients undergoing orbital ball implants after enucleation surgery with retrobulbar block alone suffered more preoperative and intraoperative anxiety，postoperative pain, and postoperative nausea and vomiting. General anesthesia alone is administered to patients undergoing orbital ball implants after enucleation surgery and opioids are used in adjunct with general anesthesia to suppress pain and hemodynamic stress associated with surgical trauma. GA only associated with more systemic opioids, short-term cognitive impairment, somnolence, and postoperative nausea and vomiting that can increase patient morbidity and delay discharge. Opioids, however, can result in adverse effects such as nausea and vomiting, pruritus, sedation. As a result of this growing demand of efficient and effective anesthesia management for orbital ball implants after enucleation surgery is becoming increasingly important. Numerous studies have reported benefits of an retrobulbar block for orbital ball implants after enucleation surgery, including quicker recovery and decreased time to discharge, decreased pain scores, opioid sparing, reduced costs, less intraoperative hemodynamic variability, improved patient satisfaction, and, in some cases, reduced GA- and/or opioid-related side effects. A recent systematic review examining all modes of postoperative pain management following orbital ball implants after enucleation surgery concluded that retrobulbar block are superior to all other forms of postoperative pain control.

DETAILED DESCRIPTION:
This retrospective review examined postoperative outcomes for orbital ball implants after enucleation surgery patients who underwent surgery with general anesthesia (GA), single-shot retrobulbar block, or retrobulbar block combined with GA. The primary outcome included postoperative pain upon arrival at and discharge from the PACU, analgesic consumption and rescue analgesia. Secondary outcomes was time to discharge from the postanesthesia care unit (PACU) as well as GA and opioid-related side effects and retrobulbar block- associated neurological complications. The investigators speculated that patients who received an retrobulbar block before GA had less postoperative pain, and reduced analgesic requirements when compared with patients who received GA Only or retrobulbar block alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they underwent orbital ball implants after enucleation surgery by one ophthalmologist surgeon specializing in oculoplastic and orbital surgery at our centre.

Exclusion Criteria:

* Patients were excluded if they underwent other concurrent surgical procedures, or were under 18 yr of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were included if they underwent orbital ball implants after enucleation surgery by one ophthalmologist surgeon specializing in oculoplastic and orbital surgery at our centre above 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2020-07-18 (Actual)

PRIMARY OUTCOMES:
postoperative pain upon arrival at and discharge from the postanesthesia care unit | through study completion: an average of 24 hour
  Visual Analogue Scale score（0-10, no pain - worse） of postoperative pain,
analgesic consumption | through study completion: an average of 24 hours
  Dose of analgesic consumption
rescue analgesia | through study completion, an average of 24 hours
  Rate of rescue analgesia

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | through study completion, an average of 24 hours
  Rate of postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Zhiying Wu, Doctor, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (2):
- China (2):
  - 叶伟娣, Hangzhou
  - Weidi Ye, Hanzhou